CLINICAL TRIAL: NCT01422954
Title: Immunization With Plasmodium Falciparum Sporozoites Under Chloroquine Versus Mefloquine Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ZonMw2
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Malaria; Plasmodium Falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Immunization; atovaquone, proguanil drug combination; Proguanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chloroquine immunisation (Active Comparator): This group will receive chloroquine prophylaxis, and three times infected mosquito-bites.
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Controlled Human Malaria Infection; Drug: Malarone
- Mefloquine immunisation (Experimental): This group will receive mefloquine prophylaxis and infected mosquito-bites.
  Interventions: Drug: Mefloquine prophylaxis; Biological: Immunization; Biological: Controlled Human Malaria Infection; Drug: Malarone
- Mefloquine control (Placebo Comparator): This group will receive mefloquine prophylaxis, and uninfected mosquito-bites.
  Interventions: Drug: Mefloquine prophylaxis; Biological: Immunization; Biological: Controlled Human Malaria Infection; Drug: Malarone

INTERVENTIONS:
Drug: Chloroquine prophylaxis — Standard prophylactic regime: a loading dose of 300 mg on day 14 and day 17 and then 300 mg once a week, starting on day 21, for a total duration of 13 weeks. On day 0, day 3, day 7 and day 10, this group will receive a placebo.
  Arms: Chloroquine immunisation
Drug: Mefloquine prophylaxis — Mefloquine prophylaxis, starting with a loading regime of split doses during the first three weeks: 125 mg on day 0, day 3, day 7, day 10, day 14 and day 17 and 250 mg once a week from day 21 onwards for a total duration of 13 weeks.
  Arms: Mefloquine control; Mefloquine immunisation
Biological: Immunization — Group 1 and 2 will receive three immunizations with Plasmodium falciparum infected mosquito-bites. Group 3 will receive an equal number of uninfected mosquito-bites.
Biological: Controlled Human Malaria Infection — Exposure to the bites of 5 Plasmodium falciparum infected mosquitoes.
Drug: Malarone — When thick smear positive, of ar day 21 after challenge, all volunteers will be treated with malarone.
  Other Names: atovaquon/proguanil

SUMMARY:
Malaria is one of the major infectious diseases in the world with a tremendous impact on the quality of life, significantly contributing to the ongoing poverty in endemic countries. It causes 800.000 deaths per year, the majority of which are children under the age of five. The malaria parasite enters the human body through the skin, by the bite of an infected mosquito. Subsequently, it invades the liver and develops and multiplies inside the hepatocytes. After a week, the hepatocytes burst open and the parasites are released in the blood stream, causing the clinical phase of the disease.

As a unique opportunity to study malaria immunology and efficacy of immunisation strategies, a protocol has been developed in the past to conduct controlled human malaria infections (CHMIs). CHMIs generally involve small groups of malaria-naïve volunteers infected via the bites of P. falciparum infected laboratory-reared Anopheline mosquitoes. Although potentially serious or even lethal, P. falciparum malaria can be radically cured at the earliest stages of blood infection when risks of complications are virtually absent.

The investigators have shown previously that healthy human volunteers can be protected from a malaria mosquito (sporozoite) challenge by immunization with sporozoites (by mosquito bites) under chloroquine prophylaxis (CPS immunization). Interestingly, sterile protection in 100% of the human CPS immunized volunteers was achieved by a relatively miniscule dose, i.e. a total of 45 infectious mosquito bites, strikingly 20-fold more potent than the 1000 bites needed in a model using irradiated mosquitoes. One possible explanation for this efficient induction of protective immunity, is the immune modulating effect of chloroquine. The investigators aim to assess this possible immune modulating effect in CPS immunization by comparing immunization with P. falciparum sporozoites under chloroquine with immunization under mefloquine prophylaxis, which has the same antimalarial effect, but not the immune modulating effects known from chloroquine.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 35 years healthy volunteers (males or females)
2. Good health based on history and clinical examination
3. Negative pregnancy test
4. Use of adequate contraception for females
5. Signing of the informed consent form, thereby demonstrating understanding of the meaning and procedures of the study
6. Agreement to inform the general practitioner and to sign a request to release medical information concerning contra-indications for participation in the study
7. Willingness to undergo a Pf controlled infection through mosquito bites
8. Agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 after challenge till treatment is finished)
9. Reachable (24/7) by mobile phone during the whole study period
10. Available to attend all study visits
11. Agreement to refrain from blood donation to Sanquin or for other purposes, during the whole study period
12. Willingness to undergo HIV, hepatitis B and hepatitis C tests
13. Negative urine toxicology screening test at screening visit and the day before challenge
14. Willingness to take a prophylactic regime of chloroquine or mefloquine and curative regimen of Malarone®

Exclusion Criteria:

1. History of malaria
2. Plans to travel to malaria endemic areas during the study period
3. Plans to travel outside of the Netherlands during the challenge period
4. Previous participation in any malaria vaccine study and/or positive serology for Pf
5. Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
6. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
7. History of arrhythmias or prolonged QT-interval
8. Positive family history in 1st and 2nd degree relatives for cardiac events < 50 years old
9. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
10. Clinically significant abnormalities in electrocardiogram (ECG) at screening
11. Body Mass Index (BMI) below 20 or above 30 kg/m2
12. Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
13. Positive HIV, HBV or HCV tests
14. Participation in any other clinical study within 30 days prior to the onset of the study
15. Enrollment in any other clinical study during the study period
16. For women: pregnancy or lactation
17. Volunteers unable to give written informed consent
18. Volunteers unable to be closely followed for social, geographic or psychological reasons
19. History of drug or alcohol abuse interfering with normal social function
20. A history of treatment for psychiatric disease or moderate or severe psychological episode in volunteer
21. A history of convulsions in volunteer
22. Severe depression, anxiety disorder of psychosis in first or second degree family
23. Contra-indications to Malarone®, chloroquine or mefloquine including hypersensitivity or treatment taken by the volunteer that interferes with Malarone®, chloroquine or mefloquine
24. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids and oral anti-histaminic are allowed) and during the study period
25. Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
26. Co-workers or trainees of the departments of Medical Microbiology, Parasitology, or Internal Medicine of the Leiden University medical Centre
27. A history of sickle cell anemia, sickle cell trait, thalassemia, thalassemia trait or G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Duration of prepatent period after challenge infection as measured by microscopy | 21 days after challenge (day 239 of the study)

SECONDARY OUTCOMES:
Development of parasitemia as measured by PCR | 21 days after challenge (day 239 of study)
Frequency of signs or symptoms in study groups | Day 0 - day 358 of study
Cellular immune responses between study groups | Day 0 -day 358 of study
Humoral immune responses between study groups | Day 0 - 358

CONTACTS AND LOCATIONS:
Overall Officials: Leo G Visser, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands

REFERENCES:
- [Derived] Bijker EM, Schats R, Obiero JM, Behet MC, van Gemert GJ, van de Vegte-Bolmer M, Graumans W, van Lieshout L, Bastiaens GJ, Teelen K, Hermsen CC, Scholzen A, Visser LG, Sauerwein RW. Sporozoite immunization of human volunteers under mefloquine prophylaxis is safe, immunogenic and protective: a double-blind randomized controlled clinical trial. PLoS One. 2014 Nov 14;9(11):e112910. doi: 10.1371/journal.pone.0112910. eCollection 2014. PMID 25396417